CLINICAL TRIAL: NCT07014618
Title: Impact of Navigator-Assisted Hypofractionation (NAVAH) on Radiation Therapy Completion in Breast Cancer and Prostate Cancer
Brief Title: Navigator-Assisted Hypofractionation (NAVAH) on Radiation Therapy Completion in Breast Cancer and Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: Gilead Sciences (Industry); Radiation Therapy Oncology Group (Network); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: OU-SCC-NAVAH
Record Dates: First submitted 2025-05-13; First posted 2025-06-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: Native American (NA)
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consented to Study: Participants in this study may provide consent in one of three ways. Consent to participate automatically includes authorization for chart review. The most comprehensive level of consent includes participation in both pre- and post-treatment surveys and receipt of navigation services as part of the study's support interventions. Another level includes consent for chart review and survey completion but a declination of navigation services. Lastly, some participants consent only to chart review and decline participation in the surveys, which automatically excludes them from receiving navigation services.
  Interventions: Other: Pre & Post Surveys; Other: Opt Out of Questionnaire

INTERVENTIONS:
Other: Pre & Post Surveys — As part of this intervention, patients will complete a pre-treatment questionnaire at the time of consent, which can be administered in person, over the phone, or through the mHealth mobile app, based on their preference. One month after treatment, patients will complete a post-treatment questionnaire using their chosen method. At the six-month mark, patients will complete an additional post-treatment questionnaire along with the COST-Functional Assessment of Chronic Illness Therapy (COST-FACT) survey.
Other: Opt Out of Questionnaire — As part of this intervention, patients declined to participate in the optional questionnaire. However, their data will still be collected through chart review and will be compared to the data of patients who accepted both the questionnaire and navigation services.

SUMMARY:
The purpose of this clinical trial is to evaluate radiation therapy (RT) completion rates among underrepresented cancer populations using qualitative measurements. Additionally, the study aims to assess the impact of patient navigators on supporting patients through their radiation care, as well as their influence on adherence to standard of care treatment modalities.

DETAILED DESCRIPTION:
The study aims to utilize qualitative measurements, including pre- and post-treatment breast and prostate cancer surveys tailored to specific ethnic groups-Native American, African American, and Hispanic/Latino populations. In addition to these culturally relevant surveys, participants will also complete the COST-Functional Assessment of Chronic Illness Therapy (COST-FACT) score to evaluate the financial and functional impact of their cancer care experience.

Those who choose to complete the surveys will be offered navigation assistance as part of the study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed Breast or Prostate Cancer.
* Subjects must be 18 years of age or older. This study requires informed consent by the subject.
* Subjects must be of African American race, Native American race, or Hispanic ethnicity.
* Subjects scheduled to undergo RT for Cancer Treatment.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects NOT of African American race, Native American race or Hispanic ethnicity.
* Subjects WITHOUT histologically/cytologically confirmed Breast or Prostate Cancer.
* Subjects younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from underrepresented minority populations (African American, Native American, and Hispanic/Latino) are eligible to be screened for the study regardless of gender. Patients must meet the inclusion criteria before consenting to the trial.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Who Complete Radiation Therapy | 6 months
  Survey-based methods will be used to assess barriers facing under-represented minority cancer patient access to patient navigation. This study will use a patient-completed, culturally sensitive survey adapted from "Walking Forward," a patient navigator program providing culturally appropriate community education on cancer, screening and treatment, to include barriers to specific RT regimens, and concerns regarding transportation.

SECONDARY OUTCOMES:
Number of Patients Successfully Impacted by Patient Navigation on Radiation Therapy | 6 Months
  Assess the impact of patient navigation on patient access to radiation oncology care [Time Frame: Immediately following radiotherapy treatment]
  Qualitative mechanisms will be used to assess the impact of patient navigation on patient access to radiation oncology care and consequently utilization of standard of care modalities. This study will use patient-completed surveys to evaluate the impact of patient navigation on access to short-course RT by using a culturally sensitive survey adapted from "Walking Forward", a patient navigator program providing culturally appropriate community education on cancer, screening and treatmen. The feedback provided by patients on the impact of patient navigation will be compared- before and after RT, and will also be compared against feedback from patients who did not received patient navigation.
Investigate The Differences in Financial Toxicity Levels | 6 Months
  This study will use patient-completed surveys to evaluate the impact of financial hardship in African-American breast cancer patients. Patient scores from an evidence-based tool, "The COmprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy (COST-FACIT)" will be used to compare financial hardship in each group of patients with early-stage breast cancer who have received a lumpectomy. Surveys will investigate differences in financial toxicity survery scores experienced by underrepresented minorities receiving conventional versus short-course RT.

CONTACTS AND LOCATIONS:
Overall Officials: Shearwood McClelland III, MD, Principal Investigator — OU Health Stephenson Cancer Center
Locations (1):
- OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No